CLINICAL TRIAL: NCT01252329
Title: High Risk Cutaneous Squamous Cell Carcinoma Treated With Mohs Surgery Randomized to Elective Management of the Draining Lymph Nodes vs. Periodic Clinical Nodal Observation
Brief Title: Comparison of Elective Lymph Node Treatment Versus Clinical Observation in the Absence of Palpable Lymph Nodes for High Risk Skin Squamous Cell Carcinoma (SCC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, John Zitelli, John A Zitelli, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO10030462
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: High Risk Cutaneous Squamous Cell Carcinoma
Keywords: high risk cutaneous squamous cell carcinoma; selective neck dissection; elective lymph node management; clinical nodal observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elective lymph node treatment arm (Active Comparator): Patients entering this arm will undergo selective nodal dissection of the draining lymph nodes with subsequent radiation and/or chemotherapy if indicated.
  Interventions: Procedure: elective lymph node dissection
- Clinical observation arm (No Intervention): Patients who enter into this arm will undergo regular, periodic clinical nodal observation with subsequent evaluation and treatment if indicated upon discovery of a palpable lymph node.

INTERVENTIONS:
Procedure: elective lymph node dissection — This entails selective lymph node dissection in patients with negative lymph node exams. The nodes dissected are those that drain from the high risk cutaneous squamous cell cancer. Subsequent radiation and/or chemotherapy may be administered in a small percentage of subjects, depending on the result of the neck dissection.
  Arms: Elective lymph node treatment arm

SUMMARY:
This study will evaluate if there is a difference in survival between elective treatment of draining lymph nodes vs. clinical nodal observation in patients undergoing Mohs surgery for high risk skin squamous cell carcinoma of the head and neck who have a normal lymph node exam. Each treatment arm is accepted as a current standard of care, and the objective is to compare outcomes between the two arms.

DETAILED DESCRIPTION:
This is a prospective, randomized, non-blinded, controlled trial of high risk head and neck cutaneous squamous cell carcinomas which will compare specific outcomes between two treatment arms. Subjects are eligible patients who are sent to Zitelli & Brodland PC for Mohs micrographic surgery of tumors that meet our high risk criteria. These patients with clinically-negative lymph node exams will either enter into the arm of nodal observation or the arm of elective management of the neck, which is currently the standard protocol per the UPMC ENT department. The patients in the observation arm will have evaluation and treatment of their lymph nodes if an abnormality is detected clinically. The primary endpoint is disease-specific survival. Secondary endpoints will include overall and disease-free survival, complications, and quality of life measures for each arm.

ELIGIBILITY:
Inclusion Criteria: Major criterion and at least one minor criteria

* Major criterion: > 6 mm depth of invasion
* Minor criteria (one or more):
* Greater than 2cm diameter
* Recurrent (prior Mohs, wide local excision, electrodesiccation and curettage, topical imiquimod or 5 fluorouracil, cryotherapy or photodynamic therapy)
* High risk location: any portion of cutaneous lip, ear, temple, scalp
* Immunosuppressed host (organ transplant recipient or chronic lymphocytic leukemia)
* Perineural invasion (yes/no; nerve involved must be greater than 0.1mm)
* Direct involvement of subcutaneous tissue (Clark's V), muscle, cartilage,or bone

Exclusion Criteria:

* Satellite metastases
* Clinically abnormal lymph node exam
* Location other than head or neck
* Exclusively mucosal squamous cell carcinoma
* Previous head and neck radiation
* In situ disease, keratoacanthoma subtypes, metatypical or collision tumors
* Inability of subject to give written informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07-14 (Actual); Study Completion 2014-07-14 (Actual)

PRIMARY OUTCOMES:
Disease-specific survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Disease-free survival | 5 years
Complications | 5 years
  This refers to any adverse event or side effect related to any of the study interventions.
quality of life | 5 years
  This refers to quality of life measured with a standard questionnaire. The two arms will be compared with respect to their differences (if any) in quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: John A Zitelli, MD, Principal Investigator — Zitelli & Brodland PC; UPMC Departments of Dermatology and Otolaryngology; David G Brodland, MD, Principal Investigator — Zitelli & Brodland PC; UPMC Departments of Dermatology and Otolaryngology; Uma Duvvuri, MD,PhD, Principal Investigator — UPMC Department of Otolaryngology; Christine H Weinberger, MD, Principal Investigator — Zitelli & Brodland PC
Locations (2):
- United States (2):
  - UPMC Department of Otolaryngology, Pittsburgh, Pennsylvania
  - Zitelli & Brodland PC, Pittsburgh, Pennsylvania